CLINICAL TRIAL: NCT02358330
Title: Project 1: Evaluating EHR-Based Health System Modifications for the Chronic Care of Smoking
Acronym: EHR Project
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-1041 EHR; A534252 (Other: UW Madison); SMPH\MEDICINE\TOBACCO RE (Other: UW Madison)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Smoking; Nicotine Dependence; Electronic Health Records; Translational Research
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EHR Enhanced Clinic Referral: A set of standard EHR modifications will be implemented in 18 clinics as part of the MBD (multiple baseline design) experiment.The key new EHR functions that will be implemented and tested are: 1) a modified "screen for smoking sta-tus" to enhance the identification and documentation of all smokers visiting targeted primary care clinics; 2) a "Smoker Registry" to track smokers, document their receipt of treatment services, and organize direct-to-consumer communications; 3) a 1-click referral system to evidence-based smoking treat-ment with UW-CTRI case managers; 4) a closed-loop feedback feature to communicate to the clinician the fate of a referral, documenting receipt of the referral and treatment engagement; and 5) EHR-based communication options to inform smokers of treatment resources
  Interventions: Other: EHR Enhanced Clinic Intervention
- Standard care (control) clinics: 10 control clinics will also be inducted into the study. These clinics will use existing EHR resources to identify smokers (e.g., the expanded vital signs) and to document their smoking status, and then use the standard paper fax-to-quit methods to refer patients to the Wisconsin Tobacco Quit Line

INTERVENTIONS:
Other: EHR Enhanced Clinic Intervention — The clinics assigned to the experimental condition will have EHR enhancements introduced.
  Groups: EHR Enhanced Clinic Referral

SUMMARY:
Smoking is the leading preventable cause of cancer mortality in the US. Despite its profound health and economic costs, smoking treatment is infrequently provided in healthcare settings, and when provided, it is not sufficiently effective. To address this, this project will develop and evaluate more efficient electronic health record (EHR) methods to identify smokers and engage them in evidence-based treatment.

DETAILED DESCRIPTION:
Specifically, this Project will develop and test new EHR enhancements and associated healthcare practices that are designed to efficiently identify smokers and recruit them into a chronic care treatment for smoking (which will be developed and evaluated in Projects 2-4). The EHR enhancements will include: 1) smoker identification and documentation aids, 2) a "Smoker Registry" (which stores relevant data on smokers and facilitates tracking their smoking status over time), 3) a 1-click system to refer smokers to the chronic care treatment for smoking, 4) a closed-loop function to provide EHR feedback to clinicians on the outcomes of their referrals, and 5) communications resources to inform smokers of treatment options and to increase their recruitment into treatment. The effects of the EHR-based enhancements and the chronic care smoking treatment will be evaluated with a multiple baseline design involving 18 primary care clinics in three healthcare systems in Wisconsin; all participants for affiliated clinical research Projects will be recruited from these clinics. This highly innovative research will evaluate the impact of an integrated set of EHR enhancements-coupled with a chronic care approach to smoking treatment-on smoker identification, and smoking treatment referral and engagement. In addition, this research will explore factors that influence the use of EHR-based enhancements in clinics. In sum, this research will develop a set of EHR-based health system enhancements that increase both the adoption of chronic care treatment by healthcare systems and smokers' engagement in that treatment.

ELIGIBILITY:
Inclusion Criteria:

* The clinics participating in the MBD experiment will be selected based on the following criteria:

  1. Size: clinics will be fairly large, including at least 4-6 clinicians, to ensure adequate recruitment for clinical trials connected with thye EHR recruitment.
  2. Location: clinics will be concentrated in Southcentral and Southeastern Wisconsin so that case managers from UW-CTRI Madison and Milwaukee research sites can provide services at multiple clinics.
  3. Diversity: clinics from each of the two health systems will include both urban and rural locations, and at least one high- and one low-SES clinic (based on rates of Medicaid and uninsured patients).
  4. Independence: clinics will not share staff or be physically adjacent to one another to combat bleeding of interventions across clinics (see 87 for the independence requirement for MBD).
  5. All clinics will routinely collect the data that will serve as dependent variables in the MBD design (this will be universal among the three health system clinics).

Exclusion Criteria:

* Any clinic not meeting the above inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a multiple baseline design with the unit of analysis as the clinic. 20-28 clinics will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 28095 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment engagement rate among smokers at a clinic | 12 months
  Percentage of those smokers identified in a clinic who engage in smoking related treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Center for Tobacco Research and Intervention — http://www.ctri.wisc.edu/